CLINICAL TRIAL: NCT07124663
Title: The Effect of Podcast Listenings and Pregnancy School Trainings in the Antenatal Period on Breastfeeding Self-Efficacy and Infant Feeding Attitudes in the Postpartum Period
Brief Title: The Effect of Podcast and Pregnancy School Education on Breastfeeding Self-Efficacy and Infant Feeding Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Yasemin Hamlaci Baskaya, doç. dr., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07082025
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Educational Podcasts, Antenatal Classes
Keywords: Self-efficacy, Pregnant women, Breastfeeding, Podcast, Education
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- podcast group (Experimental): Podcasts covering breastfeeding and breast milk education will be prepared by the educator. The content of the training will be developed in accordance with the antenatal education curriculum provided by the Ministry of Health. Pregnant women will have unrestricted access to the podcasts, allowing them to listen at any time and as often as they wish.
  Interventions: Other: Breastfeeding education
- Antenatal classes (Experimental): Presentations covering education on healthy breast milk and breastfeeding will be prepared by the educator. The content of the training presentations will be developed in accordance with the antenatal education curriculum of the Ministry of Health. The education will be delivered face-to-face once during the third trimester by the educator at the SEAH antenatal class.
  Interventions: Other: Breastfeeding education
- Control group (No Intervention): Pregnant women assigned to this group will not receive any education; only the pregnancy identification form, the Antenatal Breastfeeding Self-Efficacy Scale, and the Infant Feeding Attitude Scale will be administered.

INTERVENTIONS:
Other: Breastfeeding education — Women will receive education on breast milk and breastfeeding during pregnancy.The education program consists of two sessions, with a total duration of 60 minutes.
  Arms: Antenatal classes; podcast group

SUMMARY:
Self-efficacy is a fundamental component for individuals to effectively manage and succeed in a given domain. In this context, breastfeeding self-efficacy is essential for the successful initiation and continuation of breastfeeding. High levels of breastfeeding self-efficacy among pregnant women facilitate adaptation to the postpartum period. Educational interventions provided during the final stages of pregnancy contribute to increased self-efficacy and promote smoother adjustment to the postpartum process. Therefore, antenatal education plays a crucial role in preparing women for the postpartum period.

Accessibility to educational programs is key to reaching a larger population of pregnant women. Antenatal classes offer rich and comprehensive content, but their in-person nature requires women to physically attend clinical settings. It is essential that educational materials are also accessible to women who are unable to attend such facilities. Podcasts, which have become a part of our daily lives in recent years, can be utilized as an educational tool during pregnancy and other life stages. Podcasts are media files distributed over the internet and playable on portable devices. The core purpose of a podcast is to provide professional audio content that can be listened to anytime, anywhere, based on the listener's preference. This makes podcast-based education a highly accessible form of learning, particularly for pregnant women who can engage with the material as often as they wish, at their convenience of time and place.

Moreover, because podcasts do not involve visual elements (e.g., video or images), they can serve as a supportive platform that women can utilize during daily activities such as housework, walking, or cooking.

When reviewing previous thesis studies related to antenatal education, it is evident that most have focused on how antenatal classes affect childbirth fear and birth outcomes. On the other hand, thesis studies involving podcasts have largely been conducted in the fields of journalism, communication sciences, advertising, education, and sociology. The inclusion of a podcast intervention group in the proposed thesis will contribute novel findings from a type of intervention that has not previously been applied in the health sciences. The fact that previous podcast-related theses were in different disciplines demonstrates that podcasts are not limited to a single field but can be effective across various domains. Therefore, using podcasts during pregnancy, examining their impact on successful breastfeeding, and comparing them with a traditionally used method constitutes the most distinctive aspect of this thesis. A review of the broader literature outside of theses shows that podcasts are indeed used in the health field, primarily as a tool for raising awareness on specific topics. However, only one study in the field of obstetrics was identified, which investigated the effects of educational podcasts on women's sense of control and satisfaction during childbirth. That particular study included only low-risk pregnant women. In light of existing literature and previously conducted theses, the planned study is believed to be a novel contribution to the field of midwifery. It offers a new perspective to the literature and addresses women's health in a holistic manner by encompassing both the pregnancy and postpartum periods. This comprehensive approach is considered one of the key strengths of the research.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women who are at least in the 28th week of gestation and have not yet given birth

Pregnant women in the podcast intervention group who confirm that they can access the provided links

Pregnant women in the antenatal class education group who are able to attend the SEAH antenatal education unit

Primigravida women (women in their first pregnancy)

Exclusion Criteria:

Pregnant women diagnosed with high-risk pregnancies

Pregnant women who do not consent to participate in the study

Pregnant women who do not have sufficient proficiency in the Turkish language

Postpartum women who experienced preterm birth

Postpartum women diagnosed with a condition that results in mother-infant separation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Antenatal Breastfeeding Self-Efficacy Scale (Short Form) | Before the intervention Two weeks after the intervention
  The Breastfeeding Self-Efficacy Scale, developed by Dennis (2003), is designed to assess a mother's confidence in her ability to breastfeed her baby (Dennis, 2003). The scale was adapted into Turkish culture by Aluş Tokat et al. (2010). It includes two subscales: "technical" and "intrapersonal thoughts." The scale is a 5-point Likert type, with responses ranging from 1 = "Not at all confident" to 5 = "Always confident." The total score ranges from a minimum of 14 to a maximum of 70. A higher score indicates a higher level of breastfeeding self-efficacy. The Cronbach's alpha value for the Turkish version of the scale was reported as 0.87 (Aluş Tokat et al., 2010).
Infant Feeding Attitude Scale | Before the intervention Two weeks after the intervention Two and four weeks after birth
  The Iowa Infant Feeding Attitude Scale (IIFAS) was developed to evaluate women's attitudes toward breastfeeding, to predict infant feeding choices, and to estimate the intended duration of breastfeeding (Mora et al., 1999). The Turkish adaptation of the scale was conducted by Ekşioğlu et al. (2016). It is a 17-item, 5-point Likert-type scale with responses ranging from 1 (strongly disagree) to 5 (strongly agree). Of the 17 items, 9 support breastfeeding, while 8 are favorable toward formula feeding. Items related to formula feeding are reverse scored (Items 1, 2, 4, 6, 8, 10, 11, 14, and 17): 1=5, 2=4, 4=2, 5=1. The total attitude score ranges from a minimum of 17 (indicating a positive attitude toward bottle feeding) to a maximum of 85 (indicating a positive attitude toward breastfeeding). The scale does not have a cut-off point; higher scores indicate a more positive attitude toward breastfeeding. The Cronbach's alpha coefficient for the Turkish version was calculated as 0.71 (Ekşio
Postnatal Breastfeeding Self-Efficacy Scale (Short Form) | Two and four weeks after birth
  The Breastfeeding Self-Efficacy Scale (BSES), designed to assess a mother's confidence in her ability to breastfeed her baby, was developed by Dennis (2003). The Turkish adaptation was conducted by Aluş Tokat et al. (2010). The scale includes two subscales: "technical" and "intrapersonal thoughts." It is a 5-point Likert-type scale with responses ranging from 1 = "Not at all confident" to 5 = "Always confident." Total scores range from a minimum of 14 to a maximum of 70, with higher scores indicating greater breastfeeding self-efficacy. The Cronbach's alpha value of the Turkish original version was found to be 0.86 (Aluş Tokat et al., 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Hamlacı Başkaya, Study Director — Sakarya University
Locations (1):
- Sakarya Training and Research Hospital, Sakarya, serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No